CLINICAL TRIAL: NCT00321529
Title: Comparison of the ProAdjuster Analysis to the Penning Method of Determining Intersegmental Motion of the Cervical Spine
Status: Completed | Type: Observational
Sponsor: Logan College of Chiropractic (Other)
Other Study IDs: 0327060002
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2007-05-24 (Estimated); Status verified 2007-05

CONDITIONS: Cervical Spine Instability
Keywords: Cervical spine instability; Penning Study

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

INTERVENTIONS:
Device: motion analysis by durometer

SUMMARY:
The purpose of this study is to determine if the ProAdjuster system of analysis can be used to determine cervical spine instability using the Penning system of radiographic marking as a standard of comparison.

DETAILED DESCRIPTION:
This study will utilize the ProAdjuster Device as a method of assessing the motion of the cervical spine in participants with instability as determined by a Penning Radiographic analysis. Only participants with existing radiographic studies will be included in the study. No additional Radiographic will be required.

ELIGIBILITY:
Inclusion Criteria: Logan student, staff, or faculty with no history of ankle injury; 2. Age 18 - 60 yoa.

Exclusion Criteria: 1. Logan student, staff, or faculty ; 2. Local infection, injury or other malignancy affecting the cervical spine; 3. Any unstable joints of the cervical spine than require immobilization ; 4. Any manipulation to cervical spine within 48 hours; 5. Pregnancy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E. Enix, DC, Principal Investigator — Logan Chiropractic College
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States